CLINICAL TRIAL: NCT00772291
Title: Chronic Pain Management After Herniorraphy:Pregabalin vs Placebo. A Double-blinded Randomised Controlled Clinical Trial.
Brief Title: Chronic Pain Management After Herniorraphy
Acronym: pregabalin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, hasan eker, Prof. Dr. J.F. Lange, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pregabalin RCT
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Pain
Keywords: inguinal; hernia; chronic; pain; pregabalin; chronic pain after inguinal herniorraphy
MeSH Terms: conditions — Chronic Pain; Hernia; Bronchiolitis Obliterans Syndrome; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- pregabalin (Active Comparator)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — pregabalin 150-600mg/day during 8 weeks
  Arms: pregabalin
Drug: placebo — placebo drug during 8 weeks
  Arms: placebo

SUMMARY:
Nowadays, chronic pain mainly as a result of iatrogenic nerve damage is generally considered as the most frequent complication after inguinal hernia surgery. The primary objective of this randomised double-blind placebo-controlled trial is to investigate whether pregabalin reduces pain in patients with chronic pain of neuropathic origin after herniorraphy.

ELIGIBILITY:
Inclusion Criteria:

1. History of unilateral inguinal herniotomy
2. Establishment of neuropathic character of chronic pain by means the LANSS painscore and DN4 score
3. Abnormal sensitivity (allodynia, dysesthesia, hypoesthesia or dysesthesia) in or around the incisional area
4. Duration pain ≥ 3 months
5. Medial or lateral inguinal hernia
6. Age ≥ 18 years
7. VAS score ≥ 40 mm on Vas scale on which they indicate 'how unpleasant or disturbing the worst pain was that they had today'
8. Grade III or IV pain and discomfort on the 4-point pain and discomfort scale
9. Informed consent (addendum V)

Exclusion Criteria:

1. Participation in another trial
2. Age < 18 years
3. Cognitive disfunction
4. Patient is unable to speak Dutch
5. Hereditary problems of galactose intolerance, Lapp lactase deficiency or glucosegalactose malabsorption
6. Patient classified as American Society of Anaesthesiologist Class 4
7. Renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
pain | 8 weeks

SECONDARY OUTCOMES:
quantitative sensory testing (QST) accuracy in testing the inguinal region | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J.F. Lange, professor, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands